CLINICAL TRIAL: NCT01168349
Title: Pharmaco-epidemiological Observational Study of the Clinical Benefit of NeoRecormon® in Cancer Patients With Anemia, According to Early Response to Treatment
Brief Title: An Observational Study of NeoRecormon (Epoetin Beta) in Cancer Patients With Anemia (FAST)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22733
Record Dates: First submitted 2010-07-21; First posted 2010-07-23 (Estimated); Results first posted 2015-10-02 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Anemia, Neoplasms
MeSH Terms: conditions — Anemia; Neoplasms | interventions — epoetin beta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort
  Interventions: Drug: epoetin beta [NeoRecormon]

INTERVENTIONS:
Drug: epoetin beta [NeoRecormon] — As prescribed by physician

SUMMARY:
This observational study will evaluate the clinical benefit of NeoRecormon (epoetin beta) in daily routine practice in cancer patients with anemia. Data will be collected from patients who are receiving chemotherapy for a solid tumor or hematological malignancy. Patients will be followed for 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Patients receiving myelosuppressive chemotherapy for a solid tumor, a hematological malignancy or an autograft for hematological malignancy
* Patients for whom treatment with epoetin beta is started at the inclusion visit
* Life expectancy >/=6 months according to the physician
* Patients accepting and able to complete a French written questionnaire about his/her professional and social activities at each visit

Exclusion Criteria:

* Patients who received erythropoiesis-stimulating agents treatment, or red blood cell transfusion within 4 weeks before enrollment
* Participation in a clinical trial in onco-hematology
* Patients with myelodysplasia
* Patients with more than one active malignancy at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anemic cancer patients receiving NeoRecormon (epoetin beta)
Sampling Method: Probability Sample
Enrollment: 1060 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Neuilly-sur-Seine, France

RESULTS

PARTICIPANT FLOW:
Groups:
- Anemic Cancer Participants (Total Participants): Anemic cancer participants on NeoRecormon® injection were observed until Week 24 to 28 or early withdrawal due to death, participants' will to end the study, lost to follow-up or other reasons. The dose and frequency of NeoRecormon® were at the discretion of treating physician.
Period: Overall Study
Arm/Group | Anemic Cancer Participants (Total Participants)
Started | 1055
Completed | 754
Not Completed | 301
Not completed — Death | 157
Not completed — Lost to Follow-up | 34
Not completed — Withdrawal by Subject | 9
Not completed — Kidney transplantation | 3
Not completed — Other | 22
Not completed — Protocol Violation | 76

BASELINE CHARACTERISTICS:
Population: Efficacy population included participants who had received at least 1 dose of NeoRecormon® injection and without inclusion or exclusion criteria violation.
Arm/Group | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 979
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 528
  Male | 451

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Early Treatment Response: Day 28 to 42
Description: Early treatment response was defined as an increase of Hemoglobin (Hb) concentration of at least 1 gram/deciliter (g/dL), 4 to 6 weeks after treatment initiation.
Time Frame: Day 28 to 42
Population: Efficacy population. Here "number of participants analyzed" included those participants who were evaluable for the outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Solid Tumor Participants: Solid tumor (breast, colorectal, lung, and ovary) participants on NeoRecormon® injection were observed until Week 24 to 28 or early withdrawal due to death, participants' will to end the study, lost to follow-up or other reasons. The dose and frequency of NeoRecormon® were at the discretion of treating physician.
- Hematological Malignancy Participants: Hematological malignancy (multiple myeloma, Chronic Lymphocytic Leukemia [CLL], and lymphoma) participants on NeoRecormon® injection were observed until Week 24 to 28 or early withdrawal due to death, participants' will to end the study, lost to follow-up or other reasons. The dose and frequency of NeoRecormon® were at the discretion of treating physician.
Arm/Group | Solid Tumor Participants | Hematological Malignancy Participants | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 403 | 209 | 612
percentage of participants | 52.4 [47.48 to 57.23] | 56.5 [49.74 to 63.18] | 53.8 [49.81 to 57.71]

2. Primary Outcome: Percentage of Participants With Early Treatment Response: Day 21 to 42
Description: Early treatment response was defined as an increase of Hb concentration of at least 1 g/dL, 3 to 6 weeks after treatment initiation.
Time Frame: Day 21 to 42
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Hematological Malignancy Participants: Hematological malignancy (multiple myeloma, CLL, and lymphoma) participants on NeoRecormon® injection were observed until Week 24 to 28 or early withdrawal due to death, participants' will to end the study, lost to follow-up or other reasons. The dose and frequency of NeoRecormon® were at the discretion of treating physician.
Arm/Group | Solid Tumor Participants | Hematological Malignancy Participants | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 519 | 262 | 781
percentage of participants | 52.4 [48.11 to 56.71] | 55.7 [49.71 to 61.74] | 53.5 [50.02 to 57.02]

3. Primary Outcome: Percentage of Participants With At Least 1 Red Blood Cell (RBC) Transfusion
Description: Participants with at least 1 RBC transfusion was assessed based on the number of participants with early response or not at Day 21 to 42. Early treatment response was defined as an increase of Hb concentration of at least 1 g/dL, 3 to 6 weeks after treatment initiation.
Time Frame: Baseline up to Week 28
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- Responders: Participants who had an increase of Hb concentration of at least 1 g/dL, 3 to 6 weeks after treatment initiation.
- Non-responders: Participants who did not have an increase of Hb concentration of at least 1 g/dL, 3 to 6 weeks after treatment initiation.
Arm/Group | Responders | Non-responders | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 418 | 363 | 781
percentage of participants | 17.2 | 31.4 | 23.8
Statistical Analysis 1: Comparison: Responders vs Non-responders; Test type: Superiority or Other; Risk Ratio (RR) = 0.55, 95% CI 2-sided [0.42 to 0.71]

4. Primary Outcome: Mean Number of RBC Transfusions
Description: Mean number of transfusion was based on the number of participants with at least 1 RBC transfusion.
Time Frame: Baseline up to Week 28
Population: Efficacy population. Here "number of participants analyzed" included those participants who were evaluable for the outcome measure without any missing data.
Measure: Mean (Standard Deviation); unit: RBC transfusions
Arm/Group | Responders | Non-responders | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 67 | 111 | 178
RBC transfusions | 1.7 (1.4) | 2.1 (1.9) | 2.0 (1.8)

5. Primary Outcome: Mean Number of RBC Units
Description: Mean number of units was based on the number of participants with at least 1 RBC transfusion.
Time Frame: Baseline up to Week 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: RBC units
Arm/Group | Responders | Non-responders | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 66 | 109 | 175
RBC units | 3.4 (2.8) | 4.3 (3.9) | 4.0 (3.5)

6. Primary Outcome: Time to First RBC Transfusions
Description: Time to first RBC transfusion was assessed based on the number of participants with early response or not at Day 21 to 42. Early treatment response was defined as an increase of Hb concentration of at least 1 g/dL, 3 to 6 weeks after treatment initiation. Kaplan-Meier estimate was used.
Time Frame: Baseline up to Week 28
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Responders | Non-responders
Number analyzed (Participants) | 418 | 363
weeks | NA [NA to NA] — Median time was not reached since there were insufficient number of participants with at least 1 RBC transfusion. | NA [NA to NA] — Median time was not reached since there were insufficient number of participants with at least 1 RBC transfusion.
Statistical Analysis 1: Comparison: Responders vs Non-responders; Test type: Superiority or Other; p < 0.0001, Log Rank

7. Primary Outcome: Karnofsky Performance Status (KPS): Baseline
Description: KPS was used to quantify participant's general well-being and activities of daily life and participants were classified based on their functional impairment. An 11-level score, KPS score ranged between 0 (death) to 100 (no evidence of disease). Higher score means higher ability to perform daily tasks. KPS was based on the number of participants with early response.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Responders | Non-responders | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 411 | 359 | 770
units on a scale | 78.5 (13.1) | 78.6 (12.3) | 78.6 (12.7)

8. Primary Outcome: KPS: Week 4 to 6
Description: as for outcome 7
Time Frame: Week 4 to 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Responders | Non-responders | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 380 | 321 | 701
units on a scale | 81.2 (14.1) | 76.7 (16.2) | 79.2 (15.3)

9. Primary Outcome: KPS: Week 12 to 16
Description: as for outcome 7
Time Frame: Week 12 to 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Responders | Non-responders | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 375 | 314 | 689
units on a scale | 78.4 (22.6) | 74.7 (24.2) | 76.7 (23.4)

10. Primary Outcome: KPS: Week 24 to 28
Description: as for outcome 7
Time Frame: Week 24 to 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Responders | Non-responders | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 301 | 260 | 561
units on a scale | 79.7 (22.1) | 75.6 (24.5) | 77.8 (23.3)

11. Primary Outcome: Percentage of Participants With Professional Activity: Baseline
Description: Percentage of participants with professional activity was assessed based on the number of participants with early response or not at Day 21 to 42. Professional activity was categorized as active; disability; no occupation; retired; sick leave; student, training; and unemployment.
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Responders | Non-responders | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 418 | 363 | 781
percentage of participants
  Active | 4.1 | 3.0 | 3.6
  Disability | 2.6 | 3.3 | 2.9
  No occupation | 6.2 | 6.3 | 6.3
  Retired | 66.3 | 65 | 65.7
  Sick leave | 18.9 | 20.1 | 19.5
  Student, training | 0.2 | 0.6 | 0.4
  Unemployment | 1.7 | 1.7 | 1.7

12. Primary Outcome: Percentage of Participants With At Least 1 Sick Leave
Description: Sick leaves was described in active participants at inclusion (professional activity: active, in sick leave or unemployed participants).
Time Frame: Week 4 Up to Week 28
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Responders | Non-responders | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 103 | 90 | 193
percentage of participants | 59.2 | 74.4 | 66.3

13. Primary Outcome: Mean Number of Days of Sick Leave
Description: as for outcome 12
Time Frame: Week 4 Up to Week 28
Population: Efficacy population. Here "number of participants analyzed" included those participants who had at least 1 sick leave without any missing data.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Responders | Non-responders | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 53 | 62 | 115
days | 89.4 (62.2) | 93.3 (61.1) | 91.5 (61.4)

14. Primary Outcome: Self-Reported Questionnaire: Percentage of Participants With Current Employment at Baseline
Description: Self-administered questionnaire, work productivity and activity impairment (WPAI) questionnaire was used to assess work and activity impairment due to anemia in cancer participants in the last 7 days. The self-administered questionnaire consisted of 6 questions. It assessed amount of absenteeism, presenteeism and daily activity impairment attributable to anemia in cancer participants. Question 1 asked participants to indicate if they were currently employed or working for pay (Yes or No). Data reported for the outcome included those who were employed.
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Responders | Non-responders | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 311 | 270 | 581
percentage of participants | 6.8 | 8.1 | 7.4

15. Primary Outcome: Self-Reported Questionnaire: Percentage of Participants With Current Employment at Week 4 to 6
Description: Self-administered questionnaire, WPAI questionnaire was used to assess work and activity impairment due to anemia in cancer participants in the last 7 days. The self-administered questionnaire consisted of 6 questions. It assessed amount of absenteeism, presenteeism and daily activity impairment attributable to anemia in cancer participants. Question 1 asked participants to indicate if they were currently employed or working for pay (Yes or No). Data reported for the outcome included those who were employed.
Time Frame: Week 4 to 6
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Responders | Non-responders | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 258 | 226 | 484
percentage of participants | 5.8 | 6.2 | 6.0

16. Primary Outcome: Self-Reported Questionnaire: Percentage of Participants With Current Employment at Week 12 to 16
Description: as for outcome 15
Time Frame: Week 12 to 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Responders | Non-responders | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 235 | 209 | 444
percentage of participants | 4.3 | 4.3 | 4.3

17. Primary Outcome: Self-Reported Questionnaire: Percentage of Participants With Current Employment at Week 24 to 28
Description: as for outcome 15
Time Frame: Week 24 to 28
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Responders | Non-responders | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 163 | 147 | 310
percentage of participants | 4.9 | 4.1 | 4.5

18. Primary Outcome: Self-Reported Questionnaire: Change From Baseline on the Impact of Health on Regular Activities at Week 4 to 6
Description: Self-administered questionnaire, WPAI questionnaire was used to assess work and activity impairment due to anemia in cancer participants in the last 7 days. The self-administered questionnaire consisted of 6 questions. It assessed amount of absenteeism, presenteeism and daily activity impairment attributable to anemia in cancer participants. Question 6 asked participants to indicate how much their anemia affected their ability to do their regular daily activities such as housework, childcare, exercising, shopping, studying and so on, in the past 7 days on a scale from 0 (no effect) to 10 (completely prevented from doing daily activities).
Time Frame: Baseline, Week 4 to 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Responders | Non-responders | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 207 | 190 | 397
units on a scale
  Baseline | 6.2 (2.4) | 6.2 (2.3) | 6.2 (2.4)
  Change at Week 4 to 6 | -1.1 (2.7) | -0.8 (2.5) | -0.9 (2.6)

19. Primary Outcome: Self-Reported Questionnaire: Change From Baseline on the Impact of Health on Regular Activities at Week 12 to 16
Description: as for outcome 18
Time Frame: Baseline, Week 12 to 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Responders | Non-responders | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 195 | 175 | 370
units on a scale
  Baseline | 6.1 (2.3) | 5.9 (2.3) | 6.0 (2.3)
  Change at Week 12 to 16 | -1.5 (2.8) | -1.3 (2.9) | -1.4 (2.9)

20. Primary Outcome: Self-Reported Questionnaire: Change From Baseline on the Impact of Health on Regular Activities at Week 24 to 28
Description: as for outcome 18
Time Frame: Baseline, Week 24 to 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Responders | Non-responders | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 125 | 115 | 240
units on a scale
  Baseline | 5.9 (2.2) | 5.7 (2.3) | 5.8 (2.2)
  Change at Week 24 to 28 | -1.5 (3.0) | -1.4 (3.1) | -1.5 (3.1)

21. Secondary Outcome: Mean Starting Dose of NeoRecormon® Injection
Description: Dose of NeoRecormon® injection was measured in international units/kilograms/weeks (IU/kg/weeks).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/kg/weeks
Arm/Group | Solid Tumor Participants | Hematological Malignancy Participants | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 665 | 296 | 961
IU/kg/weeks | 471.2 (91.2) | 447.3 (95.9) | 463.9 (93.3)

22. Secondary Outcome: Percentage of Participants With Starting Dose Between 360 and 540 IU/kg/Weeks
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Solid Tumor Participants | Hematological Malignancy Participants | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 665 | 296 | 961
percentage of participants | 69.9 | 67.6 | 69.2

23. Secondary Outcome: Percentage of Participants With Pre-specified Dose and Frequency of Injections
Description: Pre-specified doses and frequency included; 20000 IU/week - Once a week (qw), 30000 IU/week -qw, 30000 IU/week - Twice a week (tw), 30000 IU/week - Once every 2 weeks (q2w), 40000 IU/week - qw, 60000 IU/week - qw, and other. Missing data were not reported.
Time Frame: Baseline, Week 4 to 6, Week 12 to 16, Week 24 to 48
Population: Efficacy population. Here "number of participants analyzed" included those participants who were evaluable for the outcome measure and "n" included participants who were evaluable at specified time point for each arm, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Solid Tumor Participants | Hematological Malignancy Participants | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 669 | 300 | 969
percentage of participants
  Baseline: 30000 IU/weeks-qw (n=669,300,969) | 97.8 | 93.7 | 96.5
  Baseline: 20000 IU/weeks-qw (n=669,300,969) | 1.2 | 3.7 | 2.0
  Baseline: 40000 IU/weeks-qw (n=669,300,969) | 0.6 | 2.3 | 1.1
  Baseline: Other (n=669,300,969) | 0.4 | 0.3 | 0.4
  Week 4-6: 30000 IU/weeks-qw (n=494,262,756) | 94.9 | 89.7 | 93.1
  Week 4-6: 20000 IU/weeks-qw (n=494,262,756) | 1.0 | 3.1 | 1.7
  Week 4-6: 30000 IU/weeks-tw (n=494,262,756) | 1.0 | 1.5 | 1.2
  Week 4-6: 60000 IU/weeks-qw (n=494,262,756) | 1.0 | 0.8 | 0.9
  Week 4-6: 30000 IU/weeks-q2w (n=494,262,756) | 0.8 | 1.5 | 1.1
  Week 4-6: 40000 IU/weeks-qw (n=494,262,756) | 0.4 | 2.7 | 1.2
  Week 4-6: Other (n=494,262,756) | 0.8 | 0.8 | 0.8
  Week 12-16: 30000 IU/weeks-qw (n=244,163,407) | 91.4 | 84.7 | 88.7
  Week 12-16: 20000 IU/weeks-qw (n=244,163,407) | 2.5 | 2.5 | 2.5
  Week 12-16: 30000 IU/weeks-tw (n=244,163,407) | 0.0 | 3.7 | 1.5
  Week 12-16: 60000 IU/weeks-qw (n=244,163,407) | 1.2 | 1.2 | 1.2
  Week 12-16: 30000 IU/weeks-q2w (n=244,163,407) | 2.5 | 3.1 | 2.7
  Week 12-16: Other (n=244,163,407) | 2.5 | 4.9 | 3.4
  Week 24-28: 30000 IU/weeks-qw (n=119,76,195) | 89.9 | 89.5 | 89.7
  Week 24-28: 20000 IU/weeks-qw (n=119,76,195) | 2.5 | 1.3 | 2.1
  Week 24-28: 60000 IU/weeks-qw (n=119,76,195) | 1.7 | 2.6 | 2.1
  Week 24-28: 40000 IU/weeks-qw (n=119,76,195) | 0.8 | 3.9 | 2.1
  Week 24-28: Other (n=119,76,195) | 5.0 | 2.6 | 4.1

24. Secondary Outcome: Percentage of Participants With Subcutaneous (SC) Route of Administration
Time Frame: Baseline, Week 4 to 6, Week 12 to 16, Week 24 to 48
Population: as for outcome 23
Measure: Number; unit: percentage of participants
Arm/Group | Solid Tumor Participants | Hematological Malignancy Participants | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 668 | 300 | 968
percentage of participants
  Baseline (n=668,300,968) | 98.7 | 100.0 | 99.1
  Week 4-6 (n=494,262,756) | 98.8 | 100.0 | 99.2
  Week 12-16 (n=238,163,401) | 98.3 | 100.0 | 99.0
  Week 24-28 (n=116,76,192) | 98.3 | 100.0 | 99.0

25. Secondary Outcome: Percentage of Participants With NeoRecormon® SC Injections at a Weekly Dose of 30000 IU
Time Frame: Baseline up to Week 28
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Solid Tumor Participants | Hematological Malignancy Participants | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 667 | 300 | 967
percentage of participants | 86.2 | 82.7 | 85.1

26. Secondary Outcome: Percentage of Participants With Modifications of NeoRecormon® Regimen
Description: All modifications were based on the change in frequency, route of administration or dose depending on the need for treatment adjustments according to Hb concentration. Percentage of participants with at least 1 modification in NeoRecormon® regimen was reported.
Time Frame: Baseline up to Week 28
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Solid Tumor Participants | Hematological Malignancy Participants | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 670 | 300 | 970
percentage of participants | 7.2 | 12.0 | 8.7

27. Secondary Outcome: Percentage of Participants With Temporary Discontinuation From NeoRecormon® Treatment
Description: Percentage of participants with at least 1 temporary discontinuation was reported.
Time Frame: Baseline up to Week 28
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Solid Tumor Participants | Hematological Malignancy Participants | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 670 | 300 | 970
percentage of participants | 8.1 | 10.3 | 8.8

28. Secondary Outcome: Percentage of Participants With Permanent Discontinuation From NeoRecormon® Treatment
Time Frame: Baseline up to Week 4 to 6, Week 12 to 16, Week 24 to 28
Population: as for outcome 23
Measure: Number; unit: percentage of participants
Arm/Group | Solid Tumor Participants | Hematological Malignancy Participants | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 639 | 294 | 933
percentage of participants
  Baseline up to Week 4-6 (n=639,294,933) | 19.9 | 8.5 | 16.3
  Baseline up to Week 12-16 (n=582,275,857) | 54.6 | 37.1 | 49.0
  Baseline up to Week 24-28 (n=457,227,684) | 74.2 | 65.6 | 71.3

29. Secondary Outcome: Relative Percent Change in Hb Concentration From Baseline Over the Study Period
Time Frame: Baseline, Week 4 to 6, Week 12 to 16, Week 24 to 28
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Solid Tumor Participants | Hematological Malignancy Participants | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 519 | 262 | 781
percent change
  Change at Week 4-6 (n=519,262,781) | 11.3 (15.9) | 13.0 (16.0) | 11.9 (15.9)
  Change at Week 12-16 (n=501,257,758) | 15.6 (19.5) | 18.6 (20.0) | 16.6 (19.7)
  Change at Week 24-28 (n=357,195,552) | 16.6 (20.2) | 24.7 (23.4) | 19.5 (21.7)

30. Secondary Outcome: Percentage of Participants With Hb Concentration Within the Range of 10 to 12 g/dL
Time Frame: Baseline up to Week 28
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Solid Tumor Participants | Hematological Malignancy Participants | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 609 | 292 | 901
percentage of participants | 36.0 | 18.5 | 30.3

31. Secondary Outcome: Percentage of Participants With Adequate Iron Status
Description: Criteria for adequate iron status included serum ferritin greater than (>) 100 micrograms/liter (µg/L) and transferrin saturation (TSAT)> 20%.
Time Frame: Baseline, Week 4 to 6, Week 12 to 16, Week 24 to 48
Population: as for outcome 23
Measure: Number; unit: percentage of participants
Arm/Group | Solid Tumor Participants | Hematological Malignancy Participants | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 58 | 65 | 123
percentage of participants
  Baseline (n=58,65,123) | 37.9 | 47.7 | 43.1
  Week 4-6 (n=31,18,49) | 22.6 | 16.7 | 20.4
  Week 12-16 (n=24,18,42) | 25.0 | 38.9 | 31.0
  Week 24-28 (n=13,17,30) | 53.8 | 70.6 | 63.3

32. Secondary Outcome: Percentage of Participants With Vitamins Prescription
Time Frame: Week 4 to 6, Week 12 to 16, Week 24 to 48
Population: as for outcome 23
Measure: Number; unit: percentage of participants
Groups:
- Lung Cancer Participants: Lung cancer participants on NeoRecormon® injection were observed until Week 24 to 28 or early withdrawal due to death, participants' will to end the study, lost to follow-up or other reasons. The dose and frequency of NeoRecormon® were at the discretion of treating physician.
- Breast Cancer Participants: Breast cancer participants on NeoRecormon® injection were observed until Week 24 to 28 or early withdrawal due to death, participants' will to end the study, lost to follow-up or other reasons. The dose and frequency of NeoRecormon® were at the discretion of treating physician.
- Colon/Rectum Cancer Participants: Colon/rectum cancer participants on NeoRecormon® injection were observed until Week 24 to 28 or early withdrawal due to death, participants' will to end the study, lost to follow-up or other reasons. The dose and frequency of NeoRecormon® were at the discretion of treating physician.
- Ovary Cancer Participants: Ovary cancer participants on NeoRecormon® injection were observed until Week 24 to 28 or early withdrawal due to death, participants' will to end the study, lost to follow-up or other reasons. The dose and frequency of NeoRecormon® were at the discretion of treating physician.
- Multiple Myeloma Participants: Multiple myeloma participants on NeoRecormon® injection were observed until Week 24 to 28 or early withdrawal due to death, participants' will to end the study, lost to follow-up or other reasons. The dose and frequency of NeoRecormon® were at the discretion of treating physician.
- Non-Hodgkin's Lymphoma Participants: Non-Hodgkin's lymphoma participants on NeoRecormon® injection were observed until Week 24 to 28 or early withdrawal due to death, participants' will to end the study, lost to follow-up or other reasons. The dose and frequency of NeoRecormon® were at the discretion of treating physician.
- Hodgkin's Lymphoma Participants: Hodgkin's lymphoma participants on NeoRecormon® injection were observed until Week 24 to 28 or early withdrawal due to death, participants' will to end the study, lost to follow-up or other reasons. The dose and frequency of NeoRecormon® were at the discretion of treating physician.
- Chronic Lymphocytic Leukemia Participants: Chronic lymphocytic leukemia participants on NeoRecormon® injection were observed until Week 24 to 28 or early withdrawal due to death, participants' will to end the study, lost to follow-up or other reasons. The dose and frequency of NeoRecormon® were at the discretion of treating physician.
Arm/Group | Lung Cancer Participants | Breast Cancer Participants | Colon/Rectum Cancer Participants | Ovary Cancer Participants | Multiple Myeloma Participants | Non-Hodgkin's Lymphoma Participants | Hodgkin's Lymphoma Participants | Chronic Lymphocytic Leukemia Participants | Anemic Cancer Participants (Total Participants)
Number analyzed (Participants) | 230 | 132 | 153 | 86 | 72 | 158 | 23 | 30 | 884
percentage of participants
  Week 4-6 (n=217,129,142,74,63,143,23,29,820) | 12.4 | 1.6 | 0.7 | 4.1 | 3.2 | 9.8 | 17.4 | 10.3 | 6.8
  Week 12-16 (n=230,132,153,86,72,158,23,30,884) | 6.5 | 0.8 | 3.9 | 3.5 | 4.2 | 8.2 | 17.4 | 10.0 | 5.4
  Week 24-28 (n=165,114,111,72,57,127,17,21,684) | 6.1 | 0.9 | 1.8 | 2.8 | 0.0 | 3.9 | 5.9 | 9.5 | 3.4

ADVERSE EVENTS:
Time Frame: Baseline up to 28 day after last dose
Description: Safety population included participants who had received at least 1 dose of NeoRecormon® injection.
Arm/Group | Solid Tumor Participants | Hematological Malignancy Participants | Anemic Cancer Participants (Total Participants)
Serious Adverse Events (participants affected / at risk) | 6/735 | 4/319 | 10/1054
Other Adverse Events (participants affected / at risk) | 63/735 | 31/319 | 94/1054
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solid Tumor Participants (N=735) | Hematological Malignancy Participants (N=319) | Anemic Cancer Participants (Total Participants) (N=1054)
Death (General disorders) | 1 (1) | 2 (2) | 3 (3)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Solid Tumor Participants (N=735) | Hematological Malignancy Participants (N=319) | Anemic Cancer Participants (Total Participants) (N=1054)
Asthenia (General disorders) | 8/8 (9) | 3 (3) | 11 (12)
Disease progression (General disorders) | 9 (9) | 1 (1) | 10 (10)
General physical health deterioration (General disorders) | 5 (5) | 1 (1) | 6 (6)
Pyrexia (General disorders) | 2 (2) | 2 (2) | 4 (4)
Hyperthermia (General disorders) | 1 (1) | 2 (3) | 3 (4)
Malaise (General disorders) | 1 (1) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 2 (2)
Catheter thrombosis (General disorders) | 1 (1) | 0 (0) | 1 (1)
Facial pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (7) | 3 (3) | 10 (10)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 3 (4) | 9 (10)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 5 (6) | 1 (1) | 6 (7)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 1 (1) | 4 (5)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 2 (2) | 1 (2) | 3 (4)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2)
Thrombocythaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 3 (3)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
HIV infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Oral fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Tonsilitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Dysaesthesia (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2)
Ageusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Phlebitis superficial (Vascular disorders) | 1 (1) | 2 (2) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 0 (0) | 3 (3)
Phlebitis (Vascular disorders) | 2 (2) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Dermititis bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Lividity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0) | 2 (2)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Initial insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Vesical fistula (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Cholestatis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.